CLINICAL TRIAL: NCT06436339
Title: Association Between Apical Periodontitis and Psoriasis Vulgaris: a Cross-sectional Study
Brief Title: Association Between Apical Periodontitis and Psoriasis Vulgaris
Status: Completed | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Simone Grandini, Head of Department of Endodontics, Periodontology, Restorative and Paediatric Dentistry, University of Siena
Other Study IDs: PSY003
Record Dates: First submitted 2024-05-23; First posted 2024-05-31 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Apical Periodontitis
Keywords: Psoriasis vulgaris
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present cross-sectional study is to assess the presence of AP and caries in psoriasis vulgaris individuals and to examine whether these medications influence these oral conditions. Therefore, 154 patients diagnosed with psoriasis were included in the study and subjected to oral examination to assess for presence of periapical lesions and caries experience.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the prevalence of apical periodontitis (AP) and caries in subjects with psoriasis vulgaris. 152 patients with psoriasis vulgaris were included in the study. The severity and extent of psoriasis were assessed according to The Psoriasis Area Severity Index (PASI), the Body Surface Area (BSA), and the Physician's Global Assessment Scale (PGA). Periapical status was assessed through dental examination and periapical radiographs. Data regarding Periapical Index (PAI), caries experience expressed as the Decayed, Missing, Filled Teeth Index (DMFT), and psoriasis medications were recorded. A predictive logistic regression model for the presence of AP and a linear regression model were then built to relate the severity and extent of AP to the type of drug therapy taken for psoriasis and to the severity and extent of the skin disease.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70
* Ability and willingness to give written consent;
* Presence of at least 6 teeth.
* Diagnosis of Psoriasis Vulgaris
* Other systemic diseases apart from psoriasis

Exclusion Criteria:

* diagnosis of periodontitis
* inability or unwillingness to give informed consent;
* periodontal treatment within the previous 6 months;
* ongoing immunosuppressive treatments or antibiotic therapy for other systemic diseases;
* pregnant or on lactation;
* additional comorbidities
* non endodontic lesions in maxilla/mandible;
* AP diagnosed on teeth with inadequate endodontic treatments and coronal restorations

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants were recruited from a specialty outpatient dermatology clinic (Unit of Dermatology, Azienda Ospedaliero-Universitaria Senese, Siena, Italy) from February 2022 to November 2023. Patients were eligible based on the inclusion criteria. Individuals were included in the study after they read and signed the written informed consent, in accordance with the Declaration of Helsinki.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Apical Periodontitis | The time frame for this observational study is defined by the initial assessment conducted at baseline. No follow-up measurements are scheduled, and the study aims to explore associations and characteristics at a single time point
  The periapical status was investigated by palpation, percussion, thermal cold testing, and panoramic radiographs. Afterward, teeth that exhibited deep carious lesions, deep restorations, no response to pulp testing, or painful response to biting and/or percussion or palpation were suspected of AP. Those teeth underwent further periapical radiograph using the long cone paralleling technique with a film holder. AP cases were diagnosed based on the identification of at least one tooth with periapical radiolucency outpacing twice the width of the periodontal ligament space and having PAI > 2.
Periapical Index Score (PAI) | The time frame for this observational study is defined by the initial assessment conducted at baseline. No follow-up measurements are scheduled, and the study aims to explore associations and characteristics at a single time point
  Periapical health was assessed radiographically using the PAI score that was determined through visual inspection of the periapical area, assigning a numerical value based on the extent and severity of inflammation. Scores ranged from 0 to 5
The DMFT index is calculated by summing the scores for decayed (D), missing (M), and filled (F) teeth for an individual or a group of individuals | The time frame for this observational study is defined by the initial assessment conducted at baseline. No follow-up measurements are scheduled, and the study aims to explore associations and characteristics at a single time point
  The DMFT index is calculated by summing the scores for decayed (D), missing (M), and filled (F) teeth for an individual or a group of individuals

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Senese, Siena, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: Undecided
no plan to share IPD